CLINICAL TRIAL: NCT01572233
Title: Effects of Personalized Physical Activity and Psycho-Education Program on Patients With Chronic Hepatitis C Infection
Brief Title: Effects of Activity and Education Program on Patients With Chronic Hepatitis C Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201103086RC
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Hepatitis C Virus Infection, Response to Therapy of
Keywords: Fatigue,Physical Activity,Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient with HCV Infection (Experimental): Personalized Physical Activity and Psycho-Education (PPAPE) Program will be tested on this group.
  Interventions: Behavioral: Personalized Physical Activity and Psycho-Education (PPAPE) Program
- usual care (No Intervention): waiting list group with usual care

INTERVENTIONS:
Behavioral: Personalized Physical Activity and Psycho-Education (PPAPE) Program — 1. Effects of Personalized Physical Activity and Psycho-Education Program on Patients with HCV infection
  2. The third and fourth year, will be examine on the 12, 24, 36, and 48 weeks during the interferon treatment.
  Arms: Patient with HCV Infection

SUMMARY:
This 4-year project will be guided by a biobehavioral model for the study of exercise interventions in two phases with the purposes to :

1. explore the patients' physical activity preferences and develop doable activity lists during treatment period
2. examine the changes of health-related physical fitness component over interferon treatment
3. develop the Personalized Physical Activity and Psych-Education (PPAPE) Program and test its effects on decreasing fatigue, physical and psychological distress, and improving their health-related physical fitness and quality of life in patients with chronic hepatitis C receiving Interferon with Ribavirin Combination Therapy
4. evaluate the outcome of the PPAPE program on increasing adherence to therapy, the sustained virological response (SVR) in 24 weeks after the end of treatment, and the time-consuming for education program during intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Hepatitis C Infection Receiving Interferon Therapy
* Aged above 18

Exclusion Criteria:

* None

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Effects of Activity and Education Program on Patients with Chronic Hepatitis C Infection | 4-year project
  Phase I of this project, the first and second year, the measurement time will be collected on the baseline (before treatment, T0), the 8 weeks (T1), 16 weeks (T2), and 24 weeks (T3) during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-ching Shun, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan